CLINICAL TRIAL: NCT00576381
Title: The Pharmacokinetics and Pharmacodynamics of Dexmedetomidine in Neonates Following Open Heart Surgery
Brief Title: Understanding Dexmedetomidine in Neonates After Open Heart Surgery
Acronym: Dex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athena Zuppa (Other)
Responsible Party: Sponsor-Investigator, Athena Zuppa, Principal Investigator, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-4-4757; CTRC 2006; NCT00516529 (obsolete NCT alias)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Tetrology of Fallot; Heart Ventricle; Hypoplastic Left Heart
Keywords: Precedex; Open Heart Surgery; Dexmedetomidine; Sedation
MeSH Terms: conditions — Tetralogy of Fallot; Hypoplastic Left Heart Syndrome | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Neonates will be administered a single bolus dose of dexmedetomidine followed by a continuous infusion for up to 24 hours post cardiac surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dosage Level 1=0.25mcg/kg loading dose, 0.2 mcg/kg/hr infusion Dosage Level 1A= 0.35mcg/kg loading dose, 0.3 mcg/kg/hr infusion Dosage Level 2= 0.5mcg/kg loading dose, 0.4 mcg/kg/hr infusion
  Other Names: Precedex

SUMMARY:
The purpose of this study is to determine what happens to dexmedetomidine in the body after it has been given to a newborn after heart surgery. We want to learn how long the drug stays in the body, how the drug is metabolized by the body, and how well the medicine works at a particular dose or amount.

DETAILED DESCRIPTION:
This is a single center, dose escalation study of a single bolus dose of dexmedetomidine followed by a continuous infusion for up to 24 hours in neonates who are immediately post-op from cardiac surgery, and require tracheal intubation with mechanical ventilation in the post-op period.

Pediatric populations may benefit from the favorable pharmacodynamic effects of this medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be less than or equal to 1 month old.
* Postconceptual age must be > or equal to 37 weeks on the day of surgery.
* Postoperative from cardiac surgery with tracheal intubation/mechanical ventilation in the immediate post-op period.
* Planned tracheal extubation within 24 hrs post-op.
* Adequate renal function (serum creatine < or equal to 1.5mg/dL)
* Adequate liver function (ALT < or equal to 165 U/L)
* Isolated heart surgery
* Informed consent

Exclusion Criteria:

* Patients who have received another investigational drug since birth.
* Patients receiving continuous infusions of muscle relaxants in the post-op setting.
* Pateints who have a positive blood culture without a subsequent negative culture of other evidence of ongoing serious infection.
* Patients who show signs and symptoms of elevated intracranial pressure.
* Post-op hypotension defined by post conceptual age.
* Pre-existing bradycardia defined by age
* Heart block
* Weight < 2kg
* Patients who, in the opinion of the investigator, are not appropriate candidates for an investigational drug study

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felice Su, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from inpatient cardiac intensive care unit prior to open heart surgery.
Groups:
- Neonatal Dose Escalation Cohorts: Neonates will be administered a single bolus dose of dexmedetomidine followed by a continuous infusion for up to 24 hours post cardiac surgery.
  Cohort 1--0.25 mcg/kg loading dose, 0.2 mcg/kg/hr infusion Cohort 1A--0.35 mcg/kg loading dose, 0.3 mcg/kg/hr infusion Cohort 2--0.5 mcg/kg loading dose, 0.4 mcg/kg/hr infusion
Period: Overall Study
Arm/Group | Neonatal Dose Escalation Cohorts
Started | 30
Completed | 23
Not Completed | 7
Not completed — Reoperation | 3
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Groups:
- Dosing Cohorts: Neonates will be administered a single bolus dose of dexmedetomidine followed by a continuous infuusion for up to 24 hours post cardiac surgery.
  Dexmedetomidine : Dosage Level 1=0.25mcg/kg loading dose, 0.2 mcg/kg/hr infusion Dosage Level 1A= 0.35mcg/kg loading dose, 0.3 mcg/kg/hr infusion Dosage Level 2= 0.5mcg/kg loading dose, 0.4 mcg/kg/hr infusion
Arm/Group | Dosing Cohorts
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: PK Profile of Dexmedetomidine
Description: This study measured the concentration of dex in the body and used those concentrations to determine how quickly the body metabolizes and eliminates dex(concentration-time or pharmacokinetic profile).The concentration of dex in the body is determined through serial blood sampling while administering dex and following discontinuation.
Time Frame: A sparse PK sampling method was utilized. Between 6-12 PK samples were drawn : After start of infusion (0.5, 4-6, 8 hours), immediately prior to end of infusion and following end of infusion (0.25, 0.5, 1, 2-4, 6-8, 10-12 & 18hrs)
Population: Based on an estimated inter-subject variability of 50% for clearance, a sample size of 32 evaluable subjects will be sufficient to detect an 18% difference (alpha 0.05, power 0.9) in the clearance in this population (38 + 18 L/hr) versus that previously reported in the adult population (46 L/hr).
Measure: Least Squares Mean (Standard Error); unit: mL/min
Groups:
- Neonates: Neonates will be administered a single bolus dose of dexmedetomidine followed by a continuous infuusion for up to 24 hours post cardiac surgery.
  Cohort 1--0.25mcg/kg loading dose, 0.2mcg/kg/hr infusion Cohort 1A--0.35 mcg/kg loading dose, 0.3 mcg/kg/hr infusion Cohort 2--0.5 mcg/kg loading dose, 0.4 mcg/kg/hr infusion
Arm/Group | Neonates
Number analyzed (Participants) | 30
mL/min | 110 (6.24) [88 to 128]

ADVERSE EVENTS:
Arm/Group | Dosing Cohorts
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Cohorts (N=30)
Atrial ectopy (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Cohorts (N=30)
myocardial ischemia (Cardiac disorders) | 1 (1)
accelerated junctional rhythm (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes